CLINICAL TRIAL: NCT05382338
Title: A Phase 3 Study of Sodium Thiosulfate for Reduction of Cisplatin-Induced Ototoxicity in Children With Average-Risk Medulloblastoma and Reduced Therapy in Children With Medulloblastoma With Low-Risk Features
Brief Title: A Study of Treatment for Medulloblastoma Using Sodium Thiosulfate to Reduce Hearing Loss
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS2031; NCI-2022-04866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS2031 (Other: Children's Oncology Group); ACNS2031 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2022-04-15; First posted 2022-05-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Childhood Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Hearing; Evoked Potentials, Auditory, Brain Stem; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Lomustine; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; sodium thiosulfate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemoradiotherapy, maintenance) (Experimental): See Detailed Description.
  Interventions: Procedure: Audiometric Test; Procedure: Auditory Brainstem Response; Procedure: Biospecimen Collection; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Lomustine; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Sodium Thiosulfate; Other: Survey Administration; Drug: Vincristine

INTERVENTIONS:
Procedure: Audiometric Test — Ancillary studies
  Other Names: Audiometric Testing; Audiometry; Hearing Test
Procedure: Auditory Brainstem Response — Ancillary studies
  Other Names: ABR; BAEP; BAER; Brainstem Auditory Evoked Potentials; Brainstem Auditory Evoked Response
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Lomustine — Given PO
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N'-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric Acid Disodium Salt
Other: Survey Administration — Ancillary studies
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase III trial tests two hypotheses in patients with low-risk and average-risk medulloblastoma. Medulloblastoma is a type of cancer that occurs in the back of the brain. The term, risk, refers to the chance of the cancer coming back after treatment. Subjects with low-risk medulloblastoma typically have a lower chance of the cancer coming back than subjects with average-risk medulloblastoma. Although treatment for newly diagnosed average-risk and low-risk medulloblastoma is generally effective at treating the cancer, there are still concerns about the side effects of such treatment. Side effects or unintended health conditions that arise due to treatment include learning difficulties, hearing loss or other issues in performing daily activities. Standard therapy for newly diagnosed average-risk or low-risk medulloblastoma includes surgery, radiation therapy, and chemotherapy (including cisplatin). Cisplatin may cause hearing loss as a side effect. In the average-risk medulloblastoma patients, this trial tests whether the addition of sodium thiosulfate (STS) to standard of care chemotherapy and radiation therapy reduces hearing loss. Previous studies with STS have shown that it may help reduce or prevent hearing loss caused by cisplatin. In the low-risk medulloblastoma patients, the study tests whether a less intense therapy (reduced radiation) can provide the same benefits as the more intense therapy. The less intense therapy may cause fewer side effects. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. The overall goals of this study are to see if giving STS along with standard treatment (radiation therapy and chemotherapy) will reduce hearing loss in medulloblastoma patients and to compare the overall outcome of patients with medulloblastoma treated with STS to patients treated without STS on a previous study in order to make sure that survival and recurrence of tumor is not worsened.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of sodium thiosulfate (STS) infusion administered during cisplatin-containing chemotherapy cycles (compared to a historical cohort selected from ACNS0331 which received chemotherapy without STS) in reducing hearing loss in children with newly-diagnosed average-risk medulloblastoma.

II. To estimate and monitor event-free survival (EFS) in this study against a carefully selected cohort from ACNS0331 to guard against loss of efficacy due to STS.

SECONDARY OBJECTIVES:

I. To estimate and monitor overall survival (OS) in this study against a carefully selected control cohort from ACNS0331.

II. To estimate the incidence of ototoxicity-related cisplatin dose modifications in the average-risk cohort.

III. To estimate the incidence of cisplatin-related nephrotoxicity in both the average-risk and low-risk cohorts.

IV. To evaluate full scale intelligence neurocognitive outcomes and trajectories of patients with average-risk medulloblastoma treated with STS compared to the control cohort from ACNS0331.

V. To evaluate quality of life and psychosocial outcomes and trajectories of patients with average-risk medulloblastoma treated with STS compared to published norms.

VI. To estimate and monitor EFS, OS, and patterns of recurrence in patients with low-risk features treated using a reduced craniospinal radiation approach.

VII. To evaluate the trajectory of hearing loss in medulloblastoma patients treated with STS.

VIII. To evaluate household material hardship as a social determinant of neurocognitive, quality of life, and psychosocial outcomes in patients with average-risk and low risk medulloblastoma.

EXPLORATORY OBJECTIVES:

I. To obtain paired blood and tumor tissue to be banked for future biology studies involving comprehensive molecular analysis, including but not limited to whole exome sequencing, ribonucleic acid (RNA) sequencing, and methylation.

II. To bank blood and cerebrospinal fluid for future studies. III. To evaluate attention, processing speed, memory, and executive function neurocognitive outcomes and trajectories, as well as hearing-related quality of life outcomes and trajectories, of patients with average-risk medulloblastoma treated with STS.

IV. To evaluate neurocognitive, quality of life, and psychosocial outcomes of patients with low-risk features treated using a reduced craniospinal radiation approach.

OUTLINE:

CHEMORADIOTHERAPY: Patients undergo radiation therapy 5 days per week for 6 weeks (weeks 1-6) and receive vincristine intravenously (IV) once weekly on weeks 2-7 in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning 4 weeks after chemoradiotherapy, patients receive lomustine orally (PO) on day 1 of cycles 1, 2, 4, 5, 7, and 8, cisplatin IV over 6 hours on day 1 of cycles 1, 2, 4, 5, 7, and 8, sodium thiosulfate IV over 15 minutes on day 1 of cycles 1, 2, 4, 5, 7, and 8, and cyclophosphamide IV over 30-60 minutes on days 1 and 2 of cycles 3, 6, and 9. Patients also receive vincristine IV on days 1, 8, and 15 of cycles 1, 2, 4, 5, 7, and 8, and on days 1 and 8 of cycles 3, 6, and 9. Treatment repeats every 6 weeks (cycles 1, 2, 4, 5, 7 and 8) or every 4 weeks (cycles 3, 6, and 9) for up to 9 cycles in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo magnetic resonance imaging (MRI) and collection of cerebrospinal fluid (CSF) throughout the study. Patients may also optionally undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for years 1-2, every 6 months for years 3-4, and then annually for years 5-10.

ELIGIBILITY:
Inclusion Criteria:

* PRE-ENROLLMENT: Patients must be ≥ 4 years and ≤ 21 years of age at the time of enrollment
* PRE-ENROLLMENT: Patient is suspected to have newly-diagnosed medulloblastoma by institutional diagnosis

  * Please note: Patients with a pending result of CSF cytology tests are eligible for NCI-2014-02057 (APEC14B1-Central Nervous System [CNS]) and CNS/Medulloblastoma Pre Enrollment Eligibility Screening
* PRE-ENROLLMENT: The patient and/or their parents or legal guardians must have signed informed consent for APEC14B1 Part A - Eligibility Screening and consent for the Molecular Characterization Initiative (MCI)
* PRE-ENROLLMENT: The required specimens are projected to be submitted under APEC14B1-CNS as soon as possible, preferably within 5 days of definitive surgery
* PRE-ENROLLMENT: All patients must have rapid central pathology review under APEC14B1-CNS prior to study enrollment on ACNS2031 step 1 in order to avoid discordant diagnoses and to verify diagnosis criterion for treatment on ACNS2031.

  * Note: Patients with a pending result of CSF cytology tests are eligible for the rapid central pathology screening review. Confirmation of CSF negativity is needed for enrollment on the ACNS2031 protocol
* PRE-ENROLLMENT: All patients must have rapid central molecular screening review under APEC14B1-CNS prior to study enrollment on ACNS2031 step 1, in order to avoid discordant diagnoses and to verify diagnosis criterion for treatment on ACNS2031
* PRE-ENROLLMENT: All patients who have histopathology confirmed must have rapid central imaging screening review under APEC14B1 prior to study enrollment on ACNS2031 step 1

  * Note: Patients must not have metastatic disease on cranial or spinal MRI. Patients with > 1.5 cm^2 residual tumor after initial surgical resection may undergo a second surgical resection prior to subsequent therapy to render them eligible for this study. The day of the second resection to remove residual tumor will be regarded as the day of definitive surgery (Day 0) and must be within a month (31 days) of the initial resection
* PRE-ENROLLMENT: All patients who have histopathology confirmed must have rapid central audiology review under APEC14B1-CNS prior to study enrollment on ACNS2031 step 1
* Patients must be >= 4 years and =< 21 years of age at the time of enrollment
* Patients must be newly diagnosed and have eligibility confirmed by rapid central pathology and molecular screening reviews performed on APEC14B1 and via the Molecular Characterization Initiative
* Average-risk cohort

  * Clinico-pathologic criteria:

    * M0 disease
    * No diffuse anaplastic histology AND
  * Molecular criteria:

    * SHH, p53wt, GLI2 normal, MYCN normal, no chromosome 14q loss
    * Group 3, MYC normal, no isochromosome 17q
    * Group 4, no chromosome 11 loss
* Low-risk features cohort

  * Clinico-pathologic criteria:

    * M0 disease
    * No diffuse anaplastic histology AND
  * Molecular criteria:

    * Group 4, chromosome 11 loss
* Patients must have negative lumbar CSF cytology

  * Note: CSF cytology for staging should be performed no sooner than 14 days post operatively to avoid false positive CSF. Ideally, CSF should be obtained between day 14 and day 21 to allow for final staging status before enrollment onto the study. Patients with positive CSF cytology obtained 0 to 14 days after surgery should have cytology repeated to determine eligibility and final CSF status. Patients with negative CSF cytology from lumbar puncture obtained 0 to 14 days after surgery do not need cytology repeated. Patients with negative CSF cytology from lumbar puncture obtained prior to surgery do not need cytology repeated post-operatively
* Patients must have eligibility confirmed by Rapid Central Imaging Review performed on APEC14B1. Patients must have =< 1.5 cm^2 cross-sectional area of residual tumor. Whole brain MRI with and without gadolinium and spine MRI with gadolinium must be performed
* Patients must weigh > 10 kg
* Patients must be enrolled, and protocol therapy must be projected to begin, no later than 31 days after definitive diagnostic surgery (day 0)
* Peripheral absolute neutrophil count (ANC) >= 1000/uL (within 7 days prior to enrollment)
* Platelet count >= 100,000/uL (transfusion independent) (within 7 days prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell count [RBC] transfusions) (within 7 days prior to enrollment)
* A serum creatinine (within 7 days prior to enrollment) based on age/sex as follows:

  * 4 to < 6 years (age); 0.8 mg/dL (male) 0.8 mg/dL (female)
  * 6 to < 10 years (age); 1 mg/dL (male) 1 mg/dL (female)
  * 10 to < 13 years (age); 1.2 mg/dL (male) 1.2 mg/dL (female)
  * 13 to < 16 years (age); 1.5 mg/dL (male) 1.4 mg/dL (female)
  * >= 16 years (age); 1.7 mg/dL (male) 1.4 mg/dL (female) OR a 24 hour urine Creatinine clearance >= 70 mL/min/1.73 m^2 (within 7 days prior to enrollment) OR a glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 (within 7 days prior to enrollment). GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)
  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Central nervous system function defined as:

  * Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
  * Patients must not be in status epilepticus, a coma or assisted ventilation at the time of study enrollment
* Auditory function defined as:

  * Patients must have normal hearing (defined as International Society of Pediatric Oncology [SIOP] grade 0) in at least one ear confirmed by rapid central audiology review performed on APEC14B1 prior to enrollment
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with metastatic disease by either MRI evaluation or lumbar CSF cytology are not eligible. Patients who are unable to undergo a lumbar puncture for assessment of CSF cytology are ineligible
* Patients must not have received any prior radiation therapy or chemotherapy (tumor-directed therapy) other than surgical intervention and/or corticosteroids
* Patients must not have any known hypersensitivity to STS, sulfates/sulfites, or other thiol agents (e.g., amifostine, n-acetylcysteine, MESNA, and captopril)
* Pregnancy and Breastfeeding:

  * Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
  * Lactating females who plan to breastfeed their infants
  * Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with >= grade 2 hearing loss | At 4 weeks after the last dose of cisplatin
  Will estimate the number and percentage of patients with >= grade 2 hearing loss using the society of pediatric oncology (SIOP) scale (defined as hearing threshold >20 dB at >= 4kHz) 4 weeks after the last dose of cisplatin. If hearing loss is observed in both ears, the worse ear will be used for this primary analysis.
Event-free survival (EFS) | From initiation of the protocol treatment to the occurrence of disease progression, disease recurrence, death from any cause, or occurrence of a second malignant neoplasm, assessed up to 10 years
  Will estimate the EFS distribution using Kaplan-Meier (KM) method.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 10 years
  Will calculate the OS distribution using KM method.
Incidence of ototoxicity-related cisplatin dose modifications in the average-risk cohort | Up to 10 years
  Will be calculated by dividing the total number of ototoxicity-related cisplatin dose modifications by the cumulative dose of cisplatin. Summary statistics including mean, standard deviation (SD), median and range will be used to summarize the data by cohorts.
Incidence of cisplatin-related nephrotoxicity in both the average-risk and low-risk cohorts | Up to 10 years
  The frequency of cisplatin-related nephrotoxicity including Grade 3 and higher creatinine increase, acute kidney injury, and chronic kidney disease will be calculated per patient as raw counts. Summary statistics will be reported including mean, median, standard deviation and range by cohorts.
Full scale intelligence neurocognitive outcomes and trajectories of patients with average-risk medulloblastoma treated with sodium thiosulfate (STS) | Up to 5 years
  A psychologist-administered battery will be used to assess longitudinal trajectories in the estimated full scale intelligence quotient (FSIQ) using the Wechsler Intelligence Scale Vocabulary and Block Design subtest. Box-plots will be drawn for each time point to visually look for change over time. Will estimate pairwise changes in FSIQ between 9 month and 30-month and between 9-month and 60-month measurements. Summary statistics will be provided for each time point and for each pairwise change including mean, standard deviation, median and range. Will compare FSIQ between two time points using parametric or non-parametric one-sample approaches depending on the normality of the data.
Quality of life and psychosocial outcomes of patients with average-risk medulloblastoma treated with STS | Up to 5 years
  Will compare quality of life (general) and psychosocial (adaptive, social, emotional, behavioral) outcomes from this study between baseline and post treatment as well as to the published healthy norms.
EFS in patients with low-risk features treated using a reduced craniospinal radiation approach | Up to 10 years
  KM estimates of the EFS distributions for the low-risk cohort will be provided.
OS in patients with low-risk features treated using a reduced craniospinal radiation approach | Up to 10 years
  KM estimates of the OS distributions for the low-risk cohort will be provided.
Patterns of recurrence in patients with low-risk features treated using a reduced craniospinal radiation approach | Up to 10 years
  The summary statistics such as count and frequency will be used to describe the patterns of recurrence.
Trajectory of hearing loss medulloblastoma patients treated with STS | Up to 60 months
  The number of patients with >= Grade 2 hearing loss using the SIOP scale in the evaluable ear at each time point will be summarized along with its 95% confidence interval.
Household material hardship as a social determinant of neurocognitive, quality of life, and psychosocial outcomes in patients with average-risk and low-risk medulloblastoma | Up to 60 months post-enrollment
  The Household Survey will be administered to parents at various timepoints to measure household material hardship. Summary statistics will be provided for each time point including mean, standard deviation, median and range for each outcome measure of interest.

OTHER OUTCOMES:
Paired blood and tumor tissue banking or future studies | Up to 5 years
  Will obtain paired blood and tumor tissue to be banked for future biology studies involving comprehensive molecular analysis.
Blood and cerebrospinal fluid banking for future studies | Up to 5 years
  Will bank blood and cerebrospinal fluid for future studies.
Attention, processing speed, memory, and executive function neurocognitive outcomes and trajectories of patients with average-risk medulloblastoma treated with STS | Up to 5 years
  Neurocognitive outcomes (attention, processing speed, and executive function) will also be examined using the approach similar to those used for FSIQ. Will be measured by the Children's Oncology Group Standardized Neuropsychological and Behavioral Batteries.
Hearing related-quality of life (HEAR-QL) of patients with average-risk medulloblastoma treated with STS | Up to 5 years
  Hearing and Audiology Survey will examine parent and patient-perceived hearing loss, hearing aid use, and barriers to hearing aid use through descriptive statistics.
HEAR-QL of patients with low-risk features treated using a reduced craniospinal radiation approach | Up to 5 years
  Hearing and Audiology Survey will examine parent and patient-perceived hearing loss, hearing aid use, and barriers to hearing aid use through descriptive statistics.
Neurocognitive, quality of life, and psychosocial outcomes of patients with low-risk features treated using a reduced craniospinal radiation approach | Up to 5 years
  The analysis approach will be similar to that for the newly diagnosed average-risk medulloblastoma. The analysis for this objective will be mainly exploratory.
Percentage of patients with >= grade 2 hearing loss in the better ear | At 4 weeks after the last dose of cisplatin
  Will report the percentage of patients with ≥ grade 2 hearing loss in the better ear at 4 weeks after the last dose of cisplatin in ACNS2031.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Salloum, Principal Investigator — Children's Oncology Group
Locations (99):
- United States (95):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - IWK Health Centre, Halifax, Nova Scotia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec